CLINICAL TRIAL: NCT02869295
Title: An Open-Label, Multicenter, Dose Escalation And Expansion Study Of NKTR-214 In Subjects With Locally Advanced Or Metastatic Solid Tumor Malignancies
Brief Title: A Phase 1/2 Multicenter Dose Escalation and Expansion Study Of NKTR-214 In Subjects With Locally Advanced Or Metastatic Solid Tumors
Acronym: NKTR-214
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-214-01; 2016-001134-10 (EudraCT Number)
Record Dates: First submitted 2016-08-03; First posted 2016-08-16 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Metastatic Solid Tumors; Locally Advanced Solid Tumors
MeSH Terms: interventions — bempegaldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NKTR-214 Dose Escalation (Experimental): This is a first in human, open-label, sequential dose escalation and expansion Phase 1 study of NKTR--214 in adult patients with locally advanced and metastatic solid tumors. The Phase 1 stage of the study is designed as an open-label dose escalation trial of NKTR--214 in participants with locally advanced or metastatic solid tumors. The goal of the dose escalation stage of the study is to find the recommended phase 2 dose, to evaluate the efficacy of NKTR--214 by assessing the objective response rate and to evaluate the safety of NKTR-214. Immunological biomarkers in plasma and tumor samples will also be measured.
  Interventions: Drug: NKTR-214

INTERVENTIONS:
Drug: NKTR-214 — Participants in the dose escalation cohorts will be treated every 21 days (q21d) or every 14 days (q14d) until tumor progression.

SUMMARY:
This is a first in human, open-label, sequential dose escalation and expansion Phase 1 study of NKTR-214 in adult patients with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a locally advanced or metastatic solid tumor.
* Received 1 or 2 prior lines of therapy.
* Life expectancy >12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Measurable disease per RECIST v1.1.
* Demonstrated adequate organ function within 14 days of treatment initiation.
* Subjects must be recovered from the effects of any prior chemotherapy, immunotherapy, other prior system anticancer therapy, radiotherapy or surgery.
* Women of childbearing potential must agree to use highly effective methods of birth control.
* All participants must agree to use double barrier contraception during study participation and for at least 2 months after the last dose of study drug.
* Additional criteria may apply.

Exclusion Criteria:

* Use of an investigational agent or an investigational device within 28 days before administration of first dose of NKTR-214.
* Females who are pregnant or breastfeeding.
* Participants who have an active autoimmune disease requiring systemic treatment within the past 3 months or have a documented history of clinically severe autoimmune disease that requires systemic steroids or immunosuppressive agents.
* Active central nervous system (CNS) metastases.
* Prior surgery or radiotherapy within 14 days of therapy.
* Participants who have had < 28 days since the last chemotherapy, immunotherapy, biological therapy, or < 14 days from approved tyrosine kinase inhibitor (TKI) therapy (sunitinib, sorafenib, vemurafenib, dabrafenib, cobimetinib), or systemic or inhaled steroid therapy at doses greater than 10mg of prednisone or equivalent before administration of the first dose of study medication.
* Participants' inability to adhere to or tolerate protocol or study procedures.
* Additional criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigator Site - New Haven, New Haven, Connecticut
  - Investigator Site - Portland, Portland, Oregon
  - Investigator Site - Houston, Houston, Texas

REFERENCES:
- [Result] Bentebibel SE, Hurwitz ME, Bernatchez C, Haymaker C, Hudgens CW, Kluger HM, Tetzlaff MT, Tagliaferri MA, Zalevsky J, Hoch U, Fanton C, Aung S, Hwu P, Curti BD, Tannir NM, Sznol M, Diab A. A First-in-Human Study and Biomarker Analysis of NKTR-214, a Novel IL2Rbetagamma-Biased Cytokine, in Patients with Advanced or Metastatic Solid Tumors. Cancer Discov. 2019 Jun;9(6):711-721. doi: 10.1158/2159-8290.CD-18-1495. Epub 2019 Apr 15. PMID 30988166
- See also: This article outlines the significance of the trial as well as the results — https://pubmed.ncbi.nlm.nih.gov/30988166/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Sponsor discontinued enrollment in order to allow the clinical development program for NKTR-214 to continue with other studies in which NKTR-214 was administered in combination with checkpoint inhibitors, based on biomarker analysis, which showed infiltration of immune cells within tumor tissue.
Groups:
- NKTR-214 0.003 mg/kg q21d: This group will be given NKTR-214 at a dose of 0.003 mg/kg every 21 days
- NKTR-214 0.006 mg/kg q21d: This group will be given NKTR-214 at a dose of 0.006 mg/kg every 21 days
- NKTR-214 0.006 mg/kg q14d: This group will be given NKTR-214 at a dose of 0.006 mg/kg every 14 days
- NKTR-214 0.009 mg/kg q21d: This group will be given NKTR-214 at a dose of 0.009 mg/kg every 21 days
- NKTR-214 0.012 mg/kg q21d: This group will be given NKTR-214 at a dose of 0.012 mg/kg every 21 days
Period: Overall Study
Arm/Group | NKTR-214 0.003 mg/kg q21d | NKTR-214 0.006 mg/kg q21d | NKTR-214 0.006 mg/kg q14d | NKTR-214 0.009 mg/kg q21d | NKTR-214 0.012 mg/kg q21d
Started | 4 | 11 | 6 | 6 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 11 | 6 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- NKTR-214 0.003 mg/kg q21d: NKTR-214 given at a dose of 0.003 mg/kg every 21 days
- NKTR-214 0.006 mg/kg q21d: NKTR-214 given at a dose of 0.006 mg/kg every 21 days
- NKTR-214 0.006 mg/kg q14d: NKTR-214 given at a dose of 0.006 mg/kg every 14 days
- NKTR-214 0.009 mg/kg q21d: NKTR-214 given at a dose of 0.009 mg/kg every 21 days
- NKTR-214 0.012 mg/kg q21d: NKTR-214 given at a dose of 0.012 mg/kg every 21 days
- Total: Total of all reporting groups
Arm/Group | NKTR-214 0.003 mg/kg q21d | NKTR-214 0.006 mg/kg q21d | NKTR-214 0.006 mg/kg q14d | NKTR-214 0.009 mg/kg q21d | NKTR-214 0.012 mg/kg q21d | Total
Number analyzed (Participants) | 4 | 11 | 6 | 6 | 1 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (14.17) | 56.5 (11.59) | 62.0 (10.16) | 60.8 (5.00) | 43.0 (NA) — There is only one participant | 57.9 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 2 | 2 | 0 | 11
  Male | 3 | 5 | 4 | 4 | 1 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 0 | 2
  White | 4 | 8 | 6 | 6 | 1 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status, n(%) [Count of Participants; unit: Participants] — GRADE - ECOG PERFORMANCE STATUS
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 3 | 7 | 2 | 3 | 1 | 16
    1 | 1 | 4 | 4 | 3 | 0 | 12
Status Enrollment [Count of Participants; unit: Participants]
  Metastatic | 4 | 9 | 6 | 6 | 1 | 26
  Locally Recurrent | 0 | 2 | 0 | 0 | 0 | 2
Lines of Prior Systemic Cancer Therapy [Mean (Standard Deviation); unit: number of lines of therapy] | 5.3 (4.72) | 1.8 (1.25) | 3.0 (2.53) | 3.3 (2.34) | 1 (NA) — Only one participant | 2.9 (2.59)
Prior Therapies [Number; unit: participants]
  # of Participants with previous Chemotherapy | 3 | 2 | 4 | 1 | 0 | 10
  # of Participants with previous Targeted Therapy | 3 | 8 | 2 | 3 | 0 | 14
  # of Participants with previous Immune Checkpoint Inhibitor (ICI) Only | 3 | 4 | 2 | 6 | 1 | 16
  # of Participants with previous ICI and other immunotherapy | 1 | 1 | 0 | 4 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Safety of NKTR-214 as Evaluated by Incidence of Drug-related Adverse Events (AEs)
Description: This outcome quantifies the number and types of adverse events associated with NKTR-214.
Time Frame: 30 days after last dose, approximately 533 days
Measure: Number; unit: events
Arm/Group | NKTR-214 0.003 mg/kg q21d | NKTR-214 0.006 mg/kg q21d | NKTR-214 0.006 mg/kg q14d | NKTR-214 0.009 mg/kg q21d | NKTR-214 0.012 mg/kg q21d
Number analyzed (Participants) | 4 | 11 | 6 | 6 | 1
events
  # of Events of Hypotension Grade 1-2 | 2 | 8 | 2 | 1 | 0
  # of Events of Syncope Grade 3-5 | 0 | 1 | 1 | 0 | 1
  # of Events of Headache Grade 1-2 | 3 | 2 | 1 | 2 | 0
  # of Events of Headache Grade 3-5 | 0 | 1 | 0 | 1 | 0
  # of Events of Anemia Grade 1-2 | 2 | 1 | 0 | 1 | 0
  # of Events of Anemia Grade 3-5 | 0 | 1 | 0 | 1 | 0
  # of Events of Metastases to Central Nervous System Grade 3-5 | 0 | 2 | 0 | 1 | 0
  # of Events of Constipation Grade 1-2 | 2 | 3 | 2 | 1 | 0
  # of Events of Constipation Grade 3-5 | 1 | 0 | 0 | 0 | 0
  # of Events of Peripheral Edema Grade 1-2 | 0 | 4 | 1 | 1 | 0
  # of Events of Peripheral Edema Grade 3-5 | 0 | 1 | 0 | 0 | 0
  # of Events of Abdominal Pain Grade 1-2 | 1 | 1 | 0 | 0 | 0
  # of Events of Abdominal pain Grade 3-5 | 0 | 0 | 2 | 0 | 0
  # of Events of Pleural Effusion Grade 1-2 | 1 | 2 | 0 | 1 | 0
  # of Events of Pleural Effusion Grade 3-5 | 1 | 0 | 0 | 0 | 0
  # of Events of Confusional State Grade 1-2 | 0 | 0 | 2 | 0 | 0
  # of Events of Confusional State Grade 3-5 | 0 | 1 | 0 | 0 | 0
  # of Events of Infusion Related Reaction Grade 1-2 | 0 | 1 | 0 | 0 | 0
  # of Events of Infusion Related Reaction Grade 3-5 | 0 | 0 | 0 | 1 | 0
  # of Events of Presyncope Grade 1-2 | 0 | 1 | 0 | 0 | 0
  # of Events of Presyncope Grade 3-5 | 0 | 1 | 0 | 0 | 0
  # of Events of Brain Edema Grade 3-5 | 0 | 1 | 0 | 0 | 0
  # of Events of Disease Progression Grade 3-5 | 0 | 0 | 1 | 0 | 0
  # of Events of Gastroduodenal Hemorrhage Grade 3-5 | 0 | 1 | 0 | 0 | 0
  # of Events of Hemiparesis Grade 3-5 | 0 | 1 | 0 | 0 | 0
  # of Events of Hypovolemic Shock Grade 3-5 | 0 | 0 | 0 | 1 | 0
  # of Events of Lipase Increased Grade 3-5 | 1 | 0 | 0 | 0 | 0
  # of Events of Liver Function Test Abnormal Grade 3-5 | 0 | 0 | 0 | 1 | 0
  # of Events of Lower Gastrointestinal Hemorrhage Grade 3-5 | 0 | 0 | 1 | 0 | 0
  # of Events of Metastases to Meninges Grade 3-5 | 0 | 1 | 0 | 0 | 0
  # of Events of Sepsis Grade 3-5 | 0 | 0 | 1 | 0 | 0
  # of Events of Fatigue Grade 1-2 | 3 | 9 | 5 | 5 | 1
  # of Events of Flu-Like Symptoms Grade 1-2 | 3 | 8 | 4 | 5 | 0
  # of Events of Pruritus Grade 1-2 | 2 | 7 | 5 | 4 | 1
  # of Events of Decreased Appetite Grade 1-2 | 1 | 6 | 4 | 4 | 0
  # of Events of Rash Grade 1-2 | 3 | 6 | 4 | 2 | 0
  # of Events of Arthralgia Grade 1-2 | 1 | 3 | 5 | 2 | 1
  # of Events of Cough Grade 1-2 | 1 | 5 | 2 | 3 | 1
  # of Events of Nausea Grade 1-2 | 3 | 3 | 3 | 2 | 0
  # of Events of Diarrhea Grade 1-2 | 3 | 2 | 1 | 3 | 0
  # of Events of Dyspnea Grade 1-2 | 3 | 4 | 1 | 0 | 0
  # of Events of Nasal Congestion Grade 1-2 | 1 | 2 | 2 | 3 | 0
  # of Events of Dizziness Grade 1-2 | 2 | 3 | 1 | 1 | 0
  # of Events of Myalgia Grade 1-2 | 0 | 3 | 1 | 2 | 0
  # of Events of Vomiting Grade 1-2 | 1 | 2 | 2 | 1 | 0
  # of Events of Weight Decreased Grade 1-2 | 2 | 1 | 0 | 2 | 0
  # of Events of Flushing Grade 1-2 | 0 | 1 | 2 | 1 | 0
  # of Event of Anxiety Grade 1-2 | 1 | 1 | 0 | 1 | 0
  # of Events of Blood creatine increased Grade 1-2 | 0 | 1 | 1 | 1 | 0
  # of Events of Cytokine Release Syndrome Grade 1-2 | 0 | 0 | 0 | 2 | 1
  # of Events of Dry Skin Grade 1-2 | 1 | 2 | 0 | 0 | 0
  # of Events of Dyspepsia Grade 1-2 | 0 | 0 | 1 | 1 | 1
  # of Events of Generalized edema Grade 1-2 | 0 | 1 | 1 | 0 | 1
  # of Events of Muscular Weakness Grade 1-2 | 1 | 1 | 1 | 0 | 0
  # of Events of Oropharyngeal Pain Grade 1-2 | 1 | 2 | 0 | 0 | 0
  # of Events of Pain Extremity Grade 1-2 | 0 | 1 | 1 | 1 | 0
  # of Events of Hypotension Grade 3-5 | 0 | 1 | 2 | 1 | 1

2. Primary Outcome: Tolerability of NKTR-214 as Evaluated by Incidence of Dose Limiting Toxicities (DLTs)
Description: The data below reflects the incidence of Dose Limiting Toxicity Events observed in this trial.
Time Frame: 30 days after last dose, up to 533 days
Measure: Number; unit: events
Arm/Group | NKTR-214 0.003 mg/kg q21d | NKTR-214 0.006 mg/kg q21d | NKTR-214 0.006 mg/kg q14d | NKTR-214 0.009 mg/kg q21d | NKTR-214 0.012 mg/kg q21d
Number analyzed (Participants) | 4 | 11 | 6 | 6 | 1
events
  # of Events of Grade 3 Hypotension | 0 | 0 | 0 | 0 | 1
  # of Events of Grade 3 Syncope | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was monitored throughout the course of the period up to 30 days after the patient received the last dose, up to 533 days.
Arm/Group | NKTR-214 0.003 mg/kg q21d | NKTR-214 0.006 mg/kg q21d | NKTR-214 0.006 mg/kg q14d | NKTR-214 0.009 mg/kg q21d | NKTR-214 0.012 mg/kg q21d
All-Cause Mortality (participants affected / at risk) | 2/4 | 3/11 | 2/6 | 1/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/4 | 5/11 | 4/6 | 3/6 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 11/11 | 6/6 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-214 0.003 mg/kg q21d (N=4) | NKTR-214 0.006 mg/kg q21d (N=11) | NKTR-214 0.006 mg/kg q14d (N=6) | NKTR-214 0.009 mg/kg q21d (N=6) | NKTR-214 0.012 mg/kg q21d (N=1)
Syncope (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Anemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Metastases to Central Nervous System (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Pain (General disorders) | 0 | 0 | 2 | 0 | 0
Ascites (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Disease Progression (General disorders) | 0 | 0 | 1 | 0 | 0
Gastroduodenal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lipase Increased (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Liver Function Test Abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 2 | 2 | 1 | 1
Cytokine Release Syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (General disorders) | 0 | 1 | 0 | 0 | 0
Humerus Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-214 0.003 mg/kg q21d (N=4) | NKTR-214 0.006 mg/kg q21d (N=11) | NKTR-214 0.006 mg/kg q14d (N=6) | NKTR-214 0.009 mg/kg q21d (N=6) | NKTR-214 0.012 mg/kg q21d (N=1)
Hypotension Grade 1-2 (Cardiac disorders) | 2 | 8 | 2 | 1 | 0
Headache Grade 1-2 (Nervous system disorders) | 3 | 2 | 1 | 2 | 0
Anemia Grade 1-2 (Cardiac disorders) | 2 | 1 | 0 | 1 | 0
Constipation Grade 1-2 (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 0
Peripheral Edema Grade 1-2 (Cardiac disorders) | 0 | 4 | 1 | 1 | 0
Abdominal Pain Grade 1-2 (General disorders) | 1 | 1 | 1 | 0 | 0
Pleural Effusion Grade 1-2 (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Confusional State Grade 1-2 (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Infusion Related Reaction Grade 1-2 (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Presyncope Grade 1-2 (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Fatigue Grade 1-2 (Cardiac disorders) | 3 | 9 | 5 | 5 | 1
Fatigue Grade 1-2 (General disorders) | 3 | 9 | 5 | 5 | 1
Flu-Like Symptoms Grade 1-2 (Infections and infestations) | 3 | 8 | 4 | 5 | 0
Pruritus Grade 1-2 (Skin and subcutaneous tissue disorders) | 2 | 7 | 5 | 4 | 1
Decreased Appetite Grade 1-2 (General disorders) | 1 | 6 | 4 | 4 | 0
Rash Grade 1-2 (Skin and subcutaneous tissue disorders) | 3 | 6 | 4 | 2 | 0
Arthralgia Grade 1-2 (General disorders) | 1 | 3 | 5 | 2 | 1
Cough Grade 1-2 (General disorders) | 1 | 5 | 2 | 3 | 1
Nausea Grade 1-2 (Gastrointestinal disorders) | 3 | 3 | 3 | 2 | 0
Diarrhea Grade 1-2 (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 0
Dyspnea Grade 1-2 (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1 | 0 | 0
Nasal Congestion Grade 1-2 (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 3 | 0
Dizziness Grade 1-2 (General disorders) | 2 | 3 | 1 | 1 | 0
Myalgia Grade 1-2 (General disorders) | 0 | 3 | 1 | 2 | 0
Vomiting Grade 1-2 (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0
Weight Decreased Grade 1-2 (General disorders) | 2 | 1 | 0 | 2 | 0
Flushing Grade 1-2 (General disorders) | 0 | 1 | 2 | 1 | 0
Anxiety Grade 1-2 (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Blood creatine increased Grade 1-2 (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Cytokine Release Syndrome Grade 1-2 (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Dry Skin Grade 1-2 (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Dyspepsia Grade 1-2 (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Generalized Edema Grade 1-2 (General disorders) | 0 | 1 | 1 | 0 | 1
Muscular Weakness Grade 1-2 (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Oropharyngeal Pain (General disorders) | 1 | 2 | 0 | 0 | 0
Pain Extremity Grade 1-2 (General disorders) | 0 | 1 | 1 | 1 | 0
Syncope Grade 3-5 (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Headache Grade 3-5 (General disorders) | 0 | 1 | 0 | 1 | 0
Anemia Grade 3-5 (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Metastases to Central Nervous System Grade 3-5 (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Constipation Grade 3-5 (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peripheral Edema Grade 3-5 (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain Grade 3-5 (General disorders) | 0 | 0 | 2 | 0 | 0
Pleural Effusion Grade 3-5 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Confusional State Grade 3-5 (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Infusion Related Reaction Grade 3-5 (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Presyncope Grade 3-5 (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Brain Edema Grade 3-5 (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Disease Progression Grade 3-5 (General disorders) | 0 | 0 | 1 | 0 | 0
Gastroduodenal Hemorrhage Grade 3-5 (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hemiparesis Grade 3-5 (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hypovolemic Shock Grade 3-5 (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Lipase Increased Grade 3-5 (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Liver Function Test Abnormal Grade 3-5 (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Lower Gastrointestinal Hemorrhage Grade 3-5 (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Metastases to Meninges Grade 3-5 (General disorders) | 0 | 1 | 0 | 0 | 0
Sepsis Grade 3-5 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypotension Grade 3-5 (Cardiac disorders) | 0 | 1 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT02869295/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT02869295/SAP_001.pdf